CLINICAL TRIAL: NCT00295685
Title: Single Dose Nexium 40MG QAM vs Lansoprazole 30mg BID for Control of Symptomatic GERD-A Double Blind Cross-Over Study
Brief Title: Nexium 40mg Once Daily vs Prevacid 30mg Twice a Day for Control of Severe GERD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Digestive & Liver Disease Specialists (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRUSESOM0159
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: GERD
Keywords: Reflux; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Antacids

INTERVENTIONS:
Drug: Antacids

SUMMARY:
The purpose of this study is to determine if people taking lansoprazole two times a day to control severe GERD symptoms can be controlled just as well, if not better, by taking Nexium just once a day.

DETAILED DESCRIPTION:
approximately 20% of patients taking first generation proton pump inhibitors (PPIs) are taking more than the standard approved dose. This dosing is required to attain adequate control of the gastric and intraesophageal pH in order to affect the desired clinical improvement. It is recognized that the b.i.d dosing strategy increases the intragastric pH control of <4 from approximately 12 hours to almost 16 hours. The refinement of the S isomer of omeprazole (Nexium)has led to a way to more effectively control acid exposure. Comparative trials with all the PPIs have shown significantly greater pH control of <4 and head to head comparisons as well as a recent crossover study. One study suggests that Nexium dosing contains approximately 16.5 hours of a pH control of <4. Conceivably, this duration of pH control suggests that b.i.d. dosing of other PPIs might be avoided. Furthermore, it suggests that patients currently taking b.i.d. PPIs might be successful candidates for conversion to q.d. Nexium. This would provide a considerable cost implication to health care plans and for patients who are responsible for paying for their PPI therapy. To date, esomeprazole has not been studied in comparison to b.i.d. dosing with other PPIs. There is pharmacologic evidence to suggest, however, that it is comparable. In this proposed study, we believe that by beginning with patients who were well controlled should make for a cleaner definition and a higher likelihood to demonstrate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of severe GERD.
* Male or female 18-80 years of age
* Ability to read, understand and provide informed consent
* GERD is Adequately controlled on BID lansoprazole as evidenced by GERD-HRQL score of </= 11
* Females of childbearing potential must use an acceptable method of birth control for the duration of the study.

Exclusion Criteria:

* Known contraindications to Nexium
* Current or historical evidence of >3 cm histologically confirmed Barrett's metaplasia without current dysplasia, esophageal stricture or extraesophageal GERD symptoms.
* Previous Esophageal gastric surgery
* Pregnant or nursing Females
* Clinically significant abnormal laboratory values
* Medical condition that may be adversely impacted by participation in this study
* History of or current drug or alcohol abuse
* Known malignancy
* Need for concurrent therapy with any acid suppressive therapy other than the study drug, antacids, alginates, NSAIDS, >165 mg ASA, prostaglandin analogs, prokinetic drug, antineoplastic agents, Ketoconazole, Itraconazole, Voriconazole, Clarithromycin, Telithromycin, HIV protease inhibitors, Rifampin, Phenobarbital, or Digoxin
* Use of investigational drug or experimental device within 30 days prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Study Completion 2007-12

PRIMARY OUTCOMES:
The proportion of subjects who are successfully stepped-down to single-dose PPI therapy, defined as having no recurrence of heartburn or acid regurgitation 3 months after PPI step-down.

SECONDARY OUTCOMES:
Changes in GERD symptom scores, health related quality of life, ancillary medication expenditures, and predictors of successful step-down.

CONTACTS AND LOCATIONS:
Overall Officials: David A Johnson, MD, Principal Investigator — Digestive & Liver Disease Specialists
Locations (1):
- Digestive & Liver Disease Specialists, Norfolk, Virginia, United States